CLINICAL TRIAL: NCT06421623
Title: Préserver Son Autonomie Par la santé du Pied : Etude d'acceptabilité d'un Programme Incluant différents Ateliers Chez Les Personnes âgées
Brief Title: Preserving Autonomy Through Foot Health: a Study on the Acceptability of a Program Including Various Workshops for the Elderly
Acronym: MINIPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH2-FUNDENBERGER-MINIPAS; 2024-A00086-41 (Other: ID-RCB)
Record Dates: First submitted 2024-03-12; First posted 2024-05-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Falling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Workshops aiming to preserve elderly's autonomy through foot health (Experimental): Study participants will benefit from a plantar massage session (5-10 min foot massage) and one posture and walking workshop per week, supervised by a trained health professional. Minimalist shoes have been purchased by the centers and used during the workshops. They will also be available to participants outside the workshops for the duration of the study.
  Interventions: Other: Program Including Various Workshops aiming to preserve elderly's autonomy through foot health

INTERVENTIONS:
Other: Program Including Various Workshops aiming to preserve elderly's autonomy through foot health — Combination of minimalist footwear, foot massages, and workshops to re-learn walking and posture

SUMMARY:
Every year in France, 2 million falls by people over 65 are responsible for 10,000 deaths, the leading cause of accidental death, and more than 130,000 hospitalizations.

The investigators will combine minimalist footwear, plantar massage, and workshops to re-learn walking and posture. The main objective of this study is to verify the acceptability and feasibility of this program among the elderly.

DETAILED DESCRIPTION:
Study participants will benefit from a plantar massage session (5-10 min massage performed by a podiatrist) and one posture and walking workshop per week, also supervised by the podiatrist. Minimalist shoes have been purchased by the centers and used during the workshops. They will also be available to participants outside the workshops for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years of age
* Able to walk independently with or without a walking aid (cane, walker, etc.)
* Persons affiliated with a social security system or assimilated
* Persons (participants, guardians, or curators where applicable) who have been informed and have given their written consent to participate in the study.

Exclusion Criteria:

* People with a contraindication to wearing minimalist shoes
* Persons unable to participate in the various workshops
* Refusal to participate in research
* Persons under court protection
* Persons unable to walk
* Persons with any other contraindication at the investigator's discretion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The acceptability of foot health workshops conducted by a podiatrist with elderly people | At the end of the 12 weeks program
  Participant acceptability will be assessed by workshop attendance rates.

SECONDARY OUTCOMES:
Foot Length measurement | Before and immediately after the intervention
  In centimeters (cm)
The distance of the center of gravity from the center | Before and immediately after the intervention
  Thanks to the stabilometry platform
Measurement of bearing surface and force distribution in static position | Before and immediately after the intervention
  Thanks to the stabilometry platform
Joint capacity for ankle flexion and extension | Before and immediately after the intervention
  Measured by the Weight-Bearing Lunge Test
Fear of falling scale | Before and immediately after the intervention
  Numerical scale from 0 to 10 (0 meaning no fear and 10 the worst fear imaginable)
The risk of falling | Before and immediately after the intervention
  Timed up and go test
Foot pain scale | Before and immediately after the intervention
  Numerical scale from 0 to 10 (0 meaning no pain and 10 the worst pain imaginable)
Number and type of foot disorders | Before and immediately after the intervention
A specifically made satisfaction questionnaire | Immediately after the intervention
  To evaluate participants' perception of the minimalist footwear and the various workshops (foot massage and walking)
Number of hours shoes used | Immediately after the intervention

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - EHPAD "Foyer Notre-Dame", Beaulieu
  - EHPAD "Vert-Bocage", Brives-Charensac
  - Ehpad Nazareth, Le Puy-en-Velay
  - Ssiad " Amadom43 ", Le Puy-en-Velay
  - EHPAD Foyer " Saint-Dominique ", Vals-près-le-Puy